CLINICAL TRIAL: NCT03411135
Title: In-depth Analysis of the Implementation of Vitiligo Extent Score (VES) Score in Comparison to Vitiligo Area and Severity Index (VASI) Score
Brief Title: Vitiligo Extent Score (VES) Score in Comparison to Vitiligo Area and Severity Index (VASI) Score
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Maha Fathy Elmasry, principal investigator, Cairo University
Other Study IDs: Dermatology6
Record Dates: First submitted 2018-01-19; First posted 2018-01-26 (Actual); Last update posted 2018-01-26 (Actual); Status verified 2018-01

CONDITIONS: Vitiligo
MeSH Terms: conditions — Vitiligo | interventions — Polyvinyl Chloride

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: VES and VASI scores as assessment methods for vitiligo — compare VES and VASI scores as assessment methods for vitiligo

SUMMARY:
All patients with vitiligo attending dermatology outpatient clinic at Kasr Alainy Teaching Hospital will be enrolled in this study to compare VES and VASI scores and evaluate them as assessment methods

ELIGIBILITY:
Inclusion Criteria:

* Age > 18.
* Non-segmental vitiligo patients

Exclusion Criteria:

* Age < 18
* Segmental vitiligo

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Vitiligo patients presenting to dermatology outpatient clinic at Kasr Alainy Teaching Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
The evaluation of the use of vitiligo extent score (VES) as a scoring system for vitiligo | 6 months